CLINICAL TRIAL: NCT02542033
Title: Double-blind, Randomized, Controlled, Cross-over Trial on Glycemic Response to Low Sugar Apple Juice
Brief Title: Glycemic Response to Low Sugar Apple Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: Nofima (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HB-RCT1-2015
Record Dates: First submitted 2015-09-03; First posted 2015-09-04 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2015-09

CONDITIONS: Impaired Fasting Glucose
Keywords: postprandial glycemia; apple juice; sugar reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- verum (Active Comparator): 500mL treated apple juice with low sugar content given on one experimental day
  Interventions: Other: treated apple juice with low sugar content
- control (Placebo Comparator): 500mL un-treated apple juice with normal sugar content given on one experimental day
  Interventions: Other: un-treated apple juice with normal sugar content

INTERVENTIONS:
Other: treated apple juice with low sugar content — Each study participant consumed 500 mL test juice at the morning of the interventional day. The 500 mL bottle content had to be ingested within 5 minutes. an intravenous catheter was inserted into a forearm vein for blood withdrawal at baseline, directly before (time point 0) and 15, 30, 45, 60, 90 and 120 minutes after starting the ingestion of the test product. From all samples plasma insulin was measured. From the blood samples taken at baseline and 120 minutes after consumption of the test product safety parameters were determined. Capillary blood was taken from the finger pad using a HemoCue® Safety Lancet at baseline (twice) and once directly before (time point 0) and 15, 30, 45, 60, 90 and 120 minutes after ingestion of the test product.
  Arms: verum
Other: un-treated apple juice with normal sugar content — Each study participant consumed 500 mL test juice at the morning of the interventional day. The 500 mL bottle content had to be ingested within 5 minutes. an intravenous catheter was inserted into a forearm vein for blood withdrawal at baseline, directly before (time point 0) and 15, 30, 45, 60, 90 and 120 minutes after starting the ingestion of the test product. From all samples plasma insulin was measured. From the blood samples taken at baseline and 120 minutes after consumption of the test product safety parameters were determined. Capillary blood was taken from the finger pad using a HemoCue® Safety Lancet at baseline (twice) and once directly before (time point 0) and 15, 30, 45, 60, 90 and 120 minutes after ingestion of the test product.
  Arms: control

SUMMARY:
Primary objective of this study is to investigate the effect of sugar reduction (starting from glucose and sucrose, respectively) on postprandial glycemic response to apple juice by comparing the reference food item apple juice (control) with the test product (apple juice with low sugar content) in male humans with impaired fasting glucose (IFG) (5.6-6.9mmol/l resp. 100-125mg/dL) (Kerner and Brückel, 2012 (DDG recommendation)) Secondary objective of this study is to investigate the effect of sugar reduction on postprandial insulinemic response.

Exploratory objectives are to investigate further characteristics of postprandial glucose and insulin response and insulin sensitivity, gastrointestinal side effects and safety aspects.

DETAILED DESCRIPTION:
Objectives:

Investigating the effect of sugar reduction in apple juice on glycemic and insulin response to ingestion of this drink.

Subjects/Methods:

In a double-blind randomized placebo-controlled clinical trial with cross-over design 30 male adults with impaired fasting glucose (IFG) received an oral drink of 500mL: 1. Verum: Apple juice, treated (low sugar content); 2. Control: Untreated apple juice (normal sugar content). Capillary blood glucose and venous plasma insulin were measured twice at baseline and then at times 0 (start of drink), 15, 30, 45, 60, 90 and 120 min.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 18y
2. diagnosed impaired fasting glucose (IFG)
3. Written informed consent

Exclusion Criteria:

1. Subjects currently enrolled in another clinical study
2. Subjects having finished another clinical study within the last 4 weeks before inclusion
3. Hypersensitivity, allergy or idiosyncratic reaction to apple, apple juice or other apple containing food
4. Acute or chronic infections
5. Renal insufficiency
6. Gastrointestinal illness
7. History of gastrointestinal surgery
8. Known fructose intolerance
9. Overt Diabetes mellitus
10. Endocrine disorders
11. Any disease or condition which might compromise significantly the hematopoietic, renal, endocrine, pulmonary, hepatic, cardiovascular, immunological, central nervous, dermatological or any other body System with the exception of the conditions defined by the inclusion criteria
12. History of hepatitis B and C
13. History of HIV infection
14. History of coagulation disorders or pharmaceutical anti-coagulation (with the exception of acetylsalicylic acid)
15. Regular medical treatment including OTC, which may have impact on the study aims (e.g. antidiabetic drugs, laxatives etc.)
16. Major cognitive or psychiatric disorders
17. Subjects who are scheduled to undergo hospitalization during the study period
18. Eating disorders (e.g. anorexia, bulimia) or special diets (e.g. vegan, vegetarian)
19. Present drug abuse or alcoholism
20. Legal incapacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
incremental area under the postprandial glucose curve | 120 min postprandially

SECONDARY OUTCOMES:
incremental area under the postprandial insulin curve | 120 min postprandially

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center (CRC) Kiel GmbH, Kiel, Schleswig-Holstein, Germany